CLINICAL TRIAL: NCT00534950
Title: Randomized Multicenter Study of 5 vs 6 Weekly Fraction of RT in the Treatment of SCC of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAC#0981-019
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2011-12

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Randomized multicenter study of 5 vs 6 weekly fraction of RT in the treatment of SCC of the head and neck
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: 5 vs 6 weekly fraction of RT — Chemotherapy

SUMMARY:
Randomized multicenter study of 5 vs 6 weekly fraction of RT in the treatment of SCC of the head and neck

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCC of the head and neck

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
safety | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Al Rajhi, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia